CLINICAL TRIAL: NCT00886158
Title: Virus Surveillance in Pediatric Solid Organ Transplant Recipients: Identifying Risk Factors for PTLD and Other Complications Post-Transplant
Brief Title: Virus Surveillance in Pediatric Solid Organ Transplant Recipients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Jodi Smith, MD, Seattle Children's Hospital
Other Study IDs: Viral PTLD
Record Dates: First submitted 2009-04-17; First posted 2009-04-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Viral Infections
Keywords: Organ Transplants
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, kidney biopsy tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Solid Organ Transplant Recipients: Solid organ transplant recipients receiving their care at Seattle Children's Hospital

SUMMARY:
Viral infections are an important complication of transplantation. Immunosuppressive therapy interferes with T cell immunity resulting in a high incidence of viral infection. Newer agents, such as mycophenolate mofetil (MMF) and sirolimus, have been associated with an increased risk of herpes virus infection. The introduction of these more potent immunosuppressive agents over the past decade correlates with an increase in the rate of hospitalizations of transplant patients with infections. This prospective study will determine the role of sub-clinical herpes virus infections in the development of complications such as chronic allograft nephropathy (CAN) and Post Transplant Lymphoproliferative Disease (PTLD). By focusing on treatable herpes virus infections, these studies have the potential to identify therapeutic strategies that can be used to diminish the burden of graft loss from CAN, significantly improving renal allograft survival and quality of life in transplant patients. Future specific interventions to test the hypothesis of a direct causal relationship between sub-clinical herpes virus infection and CAN may include the use of anti-viral therapy in response to sub-clinical infection of the renal allograft and/or peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Age from birth to 21 years
* All solid organ transplant recipients receiving their care at Seattle Children's Hospital
* Signed consent, and when age appropriate, signed assent

Exclusion Criteria:

* Lack of consent

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Solid organ transplant recipients receiving their care at Seattle Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2001-06; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate real-time quantitative PCR levels of EBV DNA for its ability to diagnose EBV infection (primary infection or reactivation), predict the development of PTLD, and compare the results to present standard of care (semi-quantitative PCR). | Specimens will be collected at the following time points post-transplant: Week 2, Week 4, Week 8, Week 10, Week 12, Month 4, Month 5, Month 6, Month 7, Month 8, Month 9, Month 10, Month 11, Month 12, Month 15, Month 18, Month 21, Month 24

SECONDARY OUTCOMES:
To describe the characteristics of EBV, CMV, HHV-6 and HHV-7 infection in the solid organ transplant population. | Specimens will be collected at the following time points post-transplant: Week 2, Week 4, Week 8, Week 10, Week 12, Month 4, Month 5, Month 6, Month 7, Month 8, Month 9, Month 10, Month 11, Month 12, Month 15, Month 18, Month 21, Month 24
To establish a tissue bank for the pediatric solid organ transplant population to allow for timely screening of this high-risk population when new technology becomes available and/or when new infectious agents are discovered | Specimens are collected at the following timepoints post transplant: 3-6 months, 12 months, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jodi Smith, MD, MPH, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States